CLINICAL TRIAL: NCT06171633
Title: Ending Sexual Harassment - Teaching Of Principal Investigators
Acronym: E-STOP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Arghavan Salles, MD, PhD, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 66842; 1R01GM147063 (NIH)
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-12

CONDITIONS: Sexual Harassment
Keywords: Sexual Harassment Prevention; Educational Online Training; Video Game Elements; Upstanding
MeSH Terms: conditions — Sexual Harassment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Intervention Group / year 1 (Experimental): Beginning in year 1, participants access online video modules through an online learning platform for up to 9 months.
  Interventions: Behavioral: E-STOP online educational program (treatment condition)
- Control Condition Group / year 1 (Experimental): Beginning in year 1, participants access online video modules through an online learning platform for up to 9 months.
  Interventions: Behavioral: E-STOP online educational program (control condition)
- Intervention Group / year 2 (Experimental): Beginning in year 2, participants access online video modules through an online learning platform for up to 9 months.
  Interventions: Behavioral: E-STOP online educational program (treatment condition)
- Control Condition Group / year 2 (Experimental): Beginning in year 2, participants access online video modules through an online learning platform for up to 9 months.
  Interventions: Behavioral: E-STOP online educational program (control condition)

INTERVENTIONS:
Behavioral: E-STOP online educational program (treatment condition) — Participants access online video modules through an online learning platform. Program includes modules on civility and upstander interventions and education about sexual harassment, microaggressions, and implicit bias.
  Arms: Intervention Group / year 1; Intervention Group / year 2
Behavioral: E-STOP online educational program (control condition) — Participants access online video modules through an online learning platform. Program includes authorship ethics only.
  Arms: Control Condition Group / year 1; Control Condition Group / year 2

SUMMARY:
The study targets three aims: Aim 1: focuses on PIs' and mentors' confidence in their ability to intervene on sexual harassment and their attitudes, perceptions, and knowledge (APK) about sexual harassment, civility, microaggressions, and unconscious bias. Aim 2: focuses on trainees' experiences of sexual harassment and microaggressions and civility, sense of belonging, well-being, productivity, and persistence in a research career. Aim 3: focuses on the culture and climate of the research learning environment.

DETAILED DESCRIPTION:
Participants (PIs, mentors, and trainees), starting in year one, will be asked to complete a baseline survey (using the secure survey software Qualtrics) regardless of condition assignment. Then, for several months, PIs, mentors, and mentees will receive virtual educational materials (presented using a Learning Management System) appropriate to the condition to which their program has been randomized.

The initial post-survey for PIs and mentors will be shortly after the final module to evaluate short-term outcomes, encompassing attitudes, perceptions, and knowledge. Subsequently, the second post-survey will be administered one year later. Trainees will participate in three post-surveys: one immediately after, another one year later, and a final one two years later.

ELIGIBILITY:
Inclusion Criteria:

* PIs, Mentors and Trainees of T-32 Programs

Exclusion Criteria:

* People who are not PIs, Mentors and Trainees of T-32 Programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2160 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Confidence to Intervene on Sexual Harassment Scale Score | Survey at baseline, immediately post-intervention (9 months after baseline), and 1 year after the completion of the 9-month intervention
  Participants are asked to rate: "How confident are you in your ability to intervene when you hear about or witness sexual harassment?" Score range: 1 (not at all confident) to 5 (extremely confident).

SECONDARY OUTCOMES:
Persistence in research careers | baseline, immediately post-intervention (9 months after baseline), and 1 year after completion of the 9-month intervention.
  Participants are asked to rate: "How extensively do you expect to be involved in research during your medical career?" Score range 1 (not involved) to 5 (exclusively)
Experiences of sexual harassment as measured by the short Sexual Experiences Questionnaire (SEQ-DoDs) | baseline, immediately post-intervention (9 months after baseline), and 1 year after completion of the 9-month intervention.
  The SEQ consists of 4 domains: gender harassment--sexist hostility (4 questions); gender harassment--sexual hostility (4 questions); unwanted sexual attention (4 questions); and sexual coercion (4 questions); the score for each question ranges from 1 (never) to 5 (many times); scores for questions within each domain are summed and divided by the number of questions, resulting in an average score range from 1 (never) to 5 (many times) for each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Arghavan Salles, Principal Investigator — arghavan@stanford.edu
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torres MB, Salles A, Cochran A. Recognizing and Reacting to Microaggressions in Medicine and Surgery. JAMA Surg. 2019 Sep 1;154(9):868-872. doi: 10.1001/jamasurg.2019.1648. PMID 31290954
- [Background] Montanaro E, Fiellin LE, Fakhouri T, Kyriakides TC, Duncan LR. Using Videogame Apps to Assess Gains in Adolescents' Substance Use Knowledge: New Opportunities for Evaluating Intervention Exposure and Content Mastery. J Med Internet Res. 2015 Oct 28;17(10):e245. doi: 10.2196/jmir.4377. PMID 26510775
- [Background] Sompayrac L, Danna KJ. An SV40 mutant oncoprotein has a nuclear location. Virology. 1989 Jul;171(1):267-70. doi: 10.1016/0042-6822(89)90536-9. PMID 2741344
- [Background] Salles A, Mueller CM, Cohen GL. Exploring the Relationship Between Stereotype Perception and Residents' Well-Being. J Am Coll Surg. 2016 Jan;222(1):52-8. doi: 10.1016/j.jamcollsurg.2015.10.004. Epub 2015 Oct 21. PMID 26616033
- [Background] Fiellin LE, Hieftje KD, Pendergrass TM, Kyriakides TC, Duncan LR, Dziura JD, Sawyer BG, Mayes L, Crusto CA, Forsyth BW, Fiellin DA. Video Game Intervention for Sexual Risk Reduction in Minority Adolescents: Randomized Controlled Trial. J Med Internet Res. 2017 Sep 18;19(9):e314. doi: 10.2196/jmir.8148. PMID 28923788
- [Background] Mueller AS, Jenkins TM, Osborne M, Dayal A, O'Connor DM, Arora VM. Gender Differences in Attending Physicians' Feedback to Residents: A Qualitative Analysis. J Grad Med Educ. 2017 Oct;9(5):577-585. doi: 10.4300/JGME-D-17-00126.1. PMID 29075375
- [Background] Tenbrunsel AE, Rees MR, Diekmann KA. Sexual Harassment in Academia: Ethical Climates and Bounded Ethicality. Annu Rev Psychol. 2019 Jan 4;70:245-270. doi: 10.1146/annurev-psych-010418-102945. Epub 2018 Aug 29. PMID 30156976
- See also: References — https://docs.google.com/document/d/1o2-5dUMHPpxm-3p3iv_6hmwRCKrlg9HK6ziX8-bN8Ow/edit